CLINICAL TRIAL: NCT02074501
Title: Supporting Older People's Informal CAREgivers at Home Through InCARE Programme
Brief Title: Intervention in Informal Caregivers Who Care Older People After a Stroke: a Pilot Study in Northern Portugal
Acronym: InCARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Minho (Other)
Responsible Party: Principal Investigator, Odete Araújo, PhD, University of Minho
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 44/2013
Record Dates: First submitted 2014-02-21; First posted 2014-02-28 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Cerebrovascular Disorder
Keywords: stroke; elderly; caregivers; empowerment; self-care; pilot study
MeSH Terms: conditions — Cerebrovascular Disorders; Stroke; Empowerment | interventions — Caregivers

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- training capacity in caregivers (Other): The participants of the InCARE programme (intervention group) will receive, additionally, intervention based on: (i) empowering caregivers to put "hands on" caring, which will be the key-point of the pilot programme; (ii) training handling techniques: mobility, bathing, (un)dressing, transferring, positioning, eating and drinking using technical aids, after 1 week, 1 month and 3 months, post hospital discharge; (iii) using telephone support, counselling caregivers on 3rd, 6th, 8th and 10th weeks post discharge. It aims at facilitating the caregivers 'adjustment to stroke demands, increasing knowledge and practical skills to support their decision-making.
  Interventions: Other: training capacity in caregivers

INTERVENTIONS:
Other: training capacity in caregivers — The participants of the InCARE programme (intervention group) will receive, additionally, intervention based on: (i) empowering caregivers to put "hands on" caring, which will be the key-point of the pilot programme; (ii) training handling techniques: mobility, bathing, (un)dressing, transferring, positioning, eating and drinking using technical aids, after 1 week, 1 month and 3 months, post hospital discharge.

SUMMARY:
Background: More than 42% of older people (aged +65) have a stroke and most of them require some type of help to self-care at home. Informal caregivers have reported different types of need and have shown dissatisfaction with technical and emotional support delivered by community health teams. Furthermore, empowering informal caregivers who care after older stroke survivors is an important challenge, preventing them from negative outcomes such as burden, anxiety and depression or loss of physical function or hospitalization in older people.

Objectives: This pilot study aims to implement and evaluate the impact of an intervention based on training and telephone support delivered to informal caregivers who care after older people post-stroke.

Setting: Community health units in Northern Portugal region. Design/Methods: This single blinded randomized trial will be delivered by a community nursing team to informal caregivers 1 week, 1 and 3 months after a hospital discharge.

Study outcome(s): The primary outcomes will be informal caregivers´ empowerment. Secondary outcomes will include burden and health quality of life in caregivers; functionality, hospital readmission and institutionalization of older people stroke survivors, measured 1 and 3 months after intervention.

Results/Conclusion: Data collection started in February and will be concluded in August 2014. First results will be published at the beginning of 2015. The InCARE programme will be the first pilot in informal caregivers study ever conducted in Portugal. It will highlight new ways to support caregivers who take care of older people after a stroke. If successful, this study will be translational and it will also allow to disseminate the results in Portugal and abroad and implement it as best practice.

DETAILED DESCRIPTION:
InCare study has a purpose to implement and evaluate an intervention delivered to informal caregivers who care for older people after a stroke.

ELIGIBILITY:
Inclusion Criteria:

Informal caregivers are eligible to participate in the InCARE programme if they meet the following inclusion criteria: (i) to be able to communicate and learn (2) not to have a cognitive disease; (3) to live in the Cávado Region covered by ACES I, II and III; (4) to return the informed consent. In addition, older stroke survivors will enter in this study if they had a stroke for the 1st time and which have become dependent for activities of daily living.

-

Exclusion Criteria:

Involvement in the InCARE programme requires to communicate frequently, face to face or on the phone, with the nursing staff. Informal caregivers will also be excluded in all the situations in which the provision of older people care is taken by formal support.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 158 (Actual)
Dates: Start 2014-01; Primary Completion 2014-02 (Actual); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Empowerment to self-care in informal caregivers | 65 years
  The primary outcomes will be informal caregivers´ empowerment to self-care. measured by ECPICID-AVC tool. This outcome will be measure 1 week and 1 month post discharge at home.
  The primary analysis will be performed according to the intention-to-treat principle.

SECONDARY OUTCOMES:
Burden | 65
  Secondary outcomes will include Burden measure by QUASCI tool in informal caregivers. This outcome will be measured 1 and 3 months after InCARE programme. All participants will be recruited through the community staff.
  This study will include a sample size of 79 informal caregivers and stroke survivors for each group.
  The descriptive statistics will describe the participants' characteristics through SPSS software.
Health quality of life | 65
  Secondary outcomes will include Health quality of life measure by SF-36 tool in informal caregivers. This outcome will be measured 1 and 3 months after InCARE programme. All participants will be recruited through the community staff.
  This study will include a sample size of 79 informal caregivers and stroke survivors for each group.
  The descriptive statistics will describe the participants' characteristics through SPSS software.

CONTACTS AND LOCATIONS:
Overall Officials: Odete Araújo, PhDs;MSc;RN, Principal Investigator — University of Minho
Locations (1):
- Odete Araújo, Braga, Norte, Portugal

REFERENCES:
- [Background] Grant JS, Elliott TR, Weaver M, Bartolucci AA, Giger JN. Telephone intervention with family caregivers of stroke survivors after rehabilitation. Stroke. 2002 Aug;33(8):2060-5. doi: 10.1161/01.str.0000020711.38824.e3. PMID 12154263
- [Background] Kalra L, Evans A, Perez I, Melbourn A, Patel A, Knapp M, Donaldson N. Training carers of stroke patients: randomised controlled trial. BMJ. 2004 May 8;328(7448):1099. doi: 10.1136/bmj.328.7448.1099. PMID 15130977
- [Background] Larson J, Franzen-Dahlin A, Billing E, Arbin M, Murray V, Wredling R. The impact of a nurse-led support and education programme for spouses of stroke patients: a randomized controlled trial. J Clin Nurs. 2005 Sep;14(8):995-1003. doi: 10.1111/j.1365-2702.2005.01206.x. PMID 16102151
- [Background] Marsden D, Quinn R, Pond N, Golledge R, Neilson C, White J, McElduff P, Pollack M. A multidisciplinary group programme in rural settings for community-dwelling chronic stroke survivors and their carers: a pilot randomized controlled trial. Clin Rehabil. 2010 Apr;24(4):328-41. doi: 10.1177/0269215509344268. Epub 2010 Feb 22. PMID 20176772
- [Background] McBride KL, White CL, Sourial R, Mayo N. Postdischarge nursing interventions for stroke survivors and their families. J Adv Nurs. 2004 Jul;47(2):192-200. doi: 10.1111/j.1365-2648.2004.03078.x. PMID 15196193
- [Background] Truelsen T, Piechowski-Jozwiak B, Bonita R, Mathers C, Bogousslavsky J, Boysen G. Stroke incidence and prevalence in Europe: a review of available data. Eur J Neurol. 2006 Jun;13(6):581-98. doi: 10.1111/j.1468-1331.2006.01138.x. PMID 16796582
- [Background] Correia M, Silva MR, Matos I, Magalhaes R, Lopes JC, Ferro JM, Silva MC. Prospective community-based study of stroke in Northern Portugal: incidence and case fatality in rural and urban populations. Stroke. 2004 Sep;35(9):2048-53. doi: 10.1161/01.STR.0000137606.34301.13. Epub 2004 Jul 15. PMID 15256683